CLINICAL TRIAL: NCT05122104
Title: Evaluation of Sarcopenia-Related Malnutrition in Older Adults According to GLIM (Global
Brief Title: Evaluation of Sarcopenia-Related Malnutrition in Older Adults
Status: Completed | Type: Observational
Sponsor: Istanbul Medeniyet University (Other)
Collaborators: Umraniye Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Esma Nur KOLBAŞI, Researcher, Istanbul Medeniyet University
Other Study IDs: IstanbulMU54
Record Dates: First submitted 2021-11-04; First posted 2021-11-16 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Sarcopenia; Malnutrition
MeSH Terms: conditions — Sarcopenia; Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Sarcopenia and malnutrition are two geriatric syndromes that are frequently seen in the elderly and have multifactorial etiology and severe clinical effects. However, the results vary widely due to the many methods and criteria used in the diagnosis and prevalence rates of both syndromes. In this study, it is aimed to investigate the relationship between the GLIM (Global Leadership Initiative on Malnutrition) criteria and various sarcopenia levels, which are newly defined worldwide and have the widest spectrum so far in describing malnutrition.

ELIGIBILITY:
Inclusion Criteria:

* To get a score of 21 and above in the Mini-Mental State Examination
* To be able to walk independently or with the help of a device (cane, etc.)

Exclusion Criteria:

* Individuals with a serious orthopedic (advanced hip or knee arthrosis, etc.) or neurologic conditions that may affect ambulation

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: community dwelling older adults
Sampling Method: Non-Probability Sample
Enrollment: 590 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-16 (Actual)

PRIMARY OUTCOMES:
Malnutrition diagnosis according to GLIM criteria | 30 minutes
  Malnutrition diagnosis according to GLIM criteria

SECONDARY OUTCOMES:
Sarcopenia diagnosis according to the European Working Group on Sarcopenia in Older People (EWGSOP) | 30 minutes
  Sarcopenia diagnosis

CONTACTS AND LOCATIONS:
Locations (1):
- Ümraniye Training and research hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Demirdag F, Kolbasi EN, Yildiz Guler K. The association between sarcopenic obesity and malnutrition in community-dwelling older adults. Age Ageing. 2025 Feb 2;54(2):afaf040. doi: 10.1093/ageing/afaf040. PMID 40036320